CLINICAL TRIAL: NCT01047553
Title: An Open Phase III, Multi-centre 52-week, Parallel-group Study Evaluating the Safety and Efficacy of Formoterol 18 μg Daily Dose Compared With Standard COPD Treatment, in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Evaluate the Safety and Efficacy of Formoterol in a Daily Dose of 18 µg (9 µg Twice Daily) in Japanese Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5122C00002
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Japanese; Phase 3; Safety; OT; Oxis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Formoterol 9 μg/dose
  Interventions: Drug: Formoterol (OT)

INTERVENTIONS:
Drug: Formoterol (OT) — 9 μg/dose, Inhaled, twice daily for 52 weeks
  Other Names: Oxis Turbuhaler®

SUMMARY:
This study is a multicentre, open, randomised, parallel-group study with formoterol 9 μg one inhalation b.i.d, or standard COPD therapy. Standard (reference) COPD treatment arm should be the group to refer to when safety results of formoterol arm will be evaluated. 240 patients with moderate-to-severe COPD will be randomised (120 patients in the formoterol-arm and 120 patients on standard COPD therapy).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, men or women ≥ 40 years
* A clinical diagnosis of COPD according to guidelines, and current COPD symptoms.
* Post-bronchodilator FEV1 < 80% of predicted normal value and FEV1/FVC < 70%, post-bronchodilator

Exclusion Criteria:

* A history and/or current clinical diagnosis of asthma and atopic diseases such as Allergic rhinitis
* Patients who have experienced COPD exacerbation requiring at least one of the following treatment, hospitalisation and/or a course of systemic steroid within 4 weeks prior to the study start.
* Significant or unstable ischaemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the investigator, or any other relevant cardiovascular disorder as judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- Japan (27):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Chitose, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Ako, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Hitachi, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kōshi, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Nagaoka, Niigata
  - Research Site, Saiki-shi, Oita Prefecture
  - Research Site, Moriguchi, Osaka
  - Research Site, Matsue, Shimane
  - Research Site, Bunkyo, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Katsushika-ku, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Tosima-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 18 December 2009, and the last participant completed the study on 20 July 2011. A total of 320 participants were enrolled at 30 centers in Japan, and 251 participants who fulfilled the randomization criteria were randomized.
Pre-assignment Details: The study started with an enrolment visit, Visit 1, 1 week prior to Visit 2, and 1 week run-in period before randomization. At Visit 2 participants had to have pre-bronchodilatory forced expiratory volume in one second (FEV1) less than 80 percent of the predicted normal value.
Groups:
- Formoterol: Formoterol 9 μg twice daily
- Standard Treatment: Standard COPD (JRS guideline and GOLD) treatment
Period: Overall Study
Arm/Group | Formoterol | Standard Treatment
Started | 125 | 126
Completed | 108 | 117
Not Completed | 17 | 9
Not completed — Adverse Event | 10 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Development of Study-Specific Withdrawal | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sever Non-Compliance to Protocol | 1 | 0
Not completed — PI's decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol | Standard Treatment | Total
Number analyzed (Participants) | 125 | 126 | 251
Age Continuous [Mean (Full Range); unit: Years] | 70.8 [43 to 88] | 70.3 [50 to 83] | 70.6 [43 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 119 | 117 | 236

OUTCOME MEASURES:

1. Primary Outcome: Clinical Laboratory Test: Haematology -Erythrocytes
Description: Mean change from Baseline
Time Frame: Baseline and week 52
Population: All randomised subjects who received at least one dose of formoterol or standard COPD treatment for each treatment group respectively and for whom any safety data after randomisation were available were included in the safety population.
Measure: Mean (Standard Deviation); unit: erythrocytes counts x10000/μl
Groups:
- Arm 1 - Formoterol: Formoterol 9 μg twice daily
- Arm 2 - Standard Treatment: Standard COPD (JRS guideline and GOLD) treatment
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
erythrocytes counts x10000/μl | -6.25 (23.8) | -5.2 (27.5)

2. Primary Outcome: Clinical Laboratory Test: Haematology -Haemoglobin
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
g/dL | -0.29 (0.73) | -0.20 (1.14)

3. Primary Outcome: Clinical Laboratory Test: Haematology-Leucocytes
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: leukocyte count/µL
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
leukocyte count/µL | -132.1 (1535.3) | -289.5 (1284.6)

4. Primary Outcome: Clinical Laboratory Test: Haematology-Platelet Count
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Platelet Count x10000/μl
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
Platelet Count x10000/μl | 0.17 (3.29) | -0.40 (4.06)

5. Primary Outcome: Clinical Laboratory Test: Haematology Eosinophils
Description: Change from baseline
Time Frame: baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Eosinophil
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of Eosinophil | 0.49 (2.21) | 0.45 (2.45)

6. Primary Outcome: Clinical Laboratory Test: Haematology Basophil
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Basophil
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of Basophil | 0.05 (0.37) | 0.01 (0.35)

7. Primary Outcome: Clinical Laboratory Test: Haematology-Lymphocytes
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Lymphocyte
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of Lymphocyte | -1.31 (7.86) | -0.43 (7.06)

8. Primary Outcome: Clinical Laboratory Test: Haematology-Monocytes
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Monocyte
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of Monocyte | -0.01 (1.55) | -0.03 (1.49)

9. Primary Outcome: Clinical Laboratory Test: Haematology -Neutrophils
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Neutrophil
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of Neutrophil | 1.92 (8.32) | -0.28 (7.64)

10. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Alanine Aminotransferase
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
U/l | -0.3 (10.0) | 4.9 (65.9)

11. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Aspartate Aminotransferase
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
U/l | 0.4 (12.0) | 2.6 (39.3)

12. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Alkaline Phosphatase (ALP)
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
U/l | 3.8 (44.7) | -4.4 (52.9)

13. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Creatinine
Description: Change from Baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mg/dL | 0.009 (0.089) | 0.021 (0.117)

14. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Total Bilirubin
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mg/dL | 0.05 (0.22) | 0.02 (0.19)

15. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Sodium
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/l
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mEq/l | -0.3 (1.9) | -0.2 (2.0)

16. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Potassium
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mEq/L | -0.15 (0.34) | -0.07 (0.37)

17. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S- Calcium
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mg/dl | -0.02 (0.42) | -0.03 (0.35)

18. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Albumin
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
g/dl | 0.00 (0.28) | 0.00 (0.23)

19. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry-S-Total Protein
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
g/dl | -0.05 (0.40) | -0.09 (0.37)

20. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry - S-Blood Urea Nitrogen (BUN)
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mg/dl | -0.48 (4.00) | 0.07 (3.99)

21. Primary Outcome: Vital Signs- Sitting SBP
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mmHg | -2.1 (14.8) | -2.1 (16.4)

22. Primary Outcome: Vital Signs- Sitting DBP
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
mmHg | -2.7 (8.9) | -3.5 (10.1)

23. Primary Outcome: Vital Signs - Pulse Rate
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
beats/minute | 1.5 (10.7) | -0.1 (10.2)

24. Primary Outcome: ECG Variables - Heart Rate
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 121 | 119
beats/min | 2.0 (11.4) | 0.6 (12.0)

25. Primary Outcome: ECG Variables - QT Interval
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milisecond
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 121 | 119
milisecond | -2.0 (22.8) | 2.6 (26.7)

26. Primary Outcome: ECG Variables - QTcB Interval
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milisecond
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 121 | 119
milisecond | 2.1 (20.6) | 1.2 (22.2)

27. Primary Outcome: ECG Variables QTcF Interval
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milisecond
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 121 | 119
milisecond | 0.5 (15.1) | 1.7 (19.1)

28. Primary Outcome: ECG Variables RR Interval
Description: Change from baseline
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milisecond
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 121 | 119
milisecond | -12.1 (7.2) | 131.7 (124.1)

29. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: The ratio of the average value of available data for mean from Weeks 0, 4, 8, 17, 26, 34, 43 and 52 to the baseline for each treatment group
Time Frame: Before randomization, 0, 4, 8, 17, 26, 34, 43 and 52 weeks after randomization
Population: All randomised subjects who received at least one dose of formoterol or standard COPD treatment for each treatment group respectively and for whom any efficacy data after randomisation were available were included in the efficacy population (Full Analysis Set: FAS).
Measure: Geometric Mean (Full Range); unit: percentage of baseline
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
percentage of baseline | 101.46 [68.9 to 139.2] | 99.42 [80.3 to 165.1]

30. Secondary Outcome: Forced Vital Capacity (FVC)
Description: The ratio of the average value of available data for Weeks 0, 4, 8, 17, 26, 34, 43 and 52 to the baseline for each treatment group
Time Frame: Before randomization, 0, 4, 8, 17, 26, 34, 43 and 52 weeks after randomization
Population: as for outcome 29
Measure: Geometric Mean (Full Range); unit: Percentage of baseline
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
Percentage of baseline | 101.62 [76.9 to 157.3] | 99.13 [75.3 to 163.0]

31. Secondary Outcome: Morning Peak Expiratory Flow(PEF)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit)and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Liter/minute (L/min)
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
Liter/minute (L/min) | 12.2 (34.9) | 7.3 (26.2)

32. Secondary Outcome: Evening Peak Expiratory Flow (PEF)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Liter/minute (L/min)
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
Liter/minute (L/min) | 9.6 (34.0) | 7.9 (28.2)

33. Secondary Outcome: Night-time Awakening Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: There are 5 alternatives (scored 0 to 4, with 4 being the most severe condition). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit ) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
units on a scale | 0.0 (0.4) | -0.1 (0.6)

34. Secondary Outcome: Daytime Breathlessness Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: as for outcome 33
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit ) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
units on a scale | -0.2 (0.7) | -0.2 (0.8)

35. Secondary Outcome: Daytime Cough Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: as for outcome 33
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
units on a scale | -0.2 (0.8) | -0.1 (0.7)

36. Secondary Outcome: Total Chronic Obstructive Pulmonary Disease (COPD) Symptom Score
Description: The Total COPD Symptom score is the sum of the measures night-time awakening, breathlessness and cough, ranges from 0 to 12 with 12 being the most severe. The change from Run-in period average to Treatment period average for each treatment group.
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit ) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
units on a scale | -0.5 (1.2) | -0.4 (1.4)

37. Secondary Outcome: Number of COPD Exacerbations Over the Treatment Period
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as worsening in COPD symptoms requiring treatment with either a course of systemic steroid or hospitalisation. Number of COPD exacerbation during 52-week randomization treatment was presented here.
Time Frame: Daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Number; unit: number of exacerbations
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
number of exacerbations | 27 | 19

38. Secondary Outcome: Use of SABA (Salbutamol) as Reliever Medication
Description: The change from Run-in period average to Treatment period average for each treatment group.
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit ) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Times/Day
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
Times/Day | -0.2 (0.7) | 0.0 (1.1)

39. Secondary Outcome: St George's Respiratory Questionnaire (SGRQ) Total Score
Description: SGRQ total score shows the impact of COPD on patient's health status, and expressed as a percentage of impairment with scale from 0 (best health status) to 100 (worst possible status). A negative rate of decline shows decreasing SGRQ total score (or improved health) over time, while a positive value shows increasing score (or worsen health). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period (14 - 18 days before Randomisation visit ) and daily during 52-week randomization treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Formoterol | Arm 2 - Standard Treatment
Number analyzed (Participants) | 125 | 126
units on a scale | -1.34 (8.48) | -0.57 (7.78)

ADVERSE EVENTS:
Arm/Group | Formoterol | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 20/125 | 18/126
Other Adverse Events (participants affected / at risk) | 54/125 | 60/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol (N=125) | Standard Treatment (N=126)
Aortic Dissection (Vascular disorders) | 1 | 0
Spermatic Cord Disorder (Reproductive system and breast disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Chest X-Ray Abnormal (Investigations) | 1 | 0
Device Failure (General disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Stomach Mass (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Lacunar Infarction (Nervous system disorders) | 0 | 1
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Brain Stem Infarction (Nervous system disorders) | 0 | 1
Venom Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Cord Injury Cervical (Injury, poisoning and procedural complications) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Squamous Cell Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Bipolar Disorder (Psychiatric disorders) | 0 | 1
SPERMATIC CORD DISORDER (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol (N=125) | Standard Treatment (N=126)
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 | 0
Influenza (Infections and infestations) | 1 | 3
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 3
Palpitations (Cardiac disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 2
Headache (Nervous system disorders) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Rhinitis (Infections and infestations) | 5 | 2
Insomnia (Psychiatric disorders) | 3 | 4
Hypertension (Vascular disorders) | 3 | 5
Gastritis (Gastrointestinal disorders) | 3 | 5
Dizziness (Nervous system disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 5 | 4
Conjunctivitis (Eye disorders) | 5 | 5
Pneumonia (Infections and infestations) | 8 | 3
Pharyngitis (Infections and infestations) | 7 | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Bronchitis (Infections and infestations) | 5 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 2
NASOPHARYNGITIS (Infections and infestations) | 42 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other